CLINICAL TRIAL: NCT06322511
Title: The Effectiveness of Dialogical Family Guidance in Families With a Child With Neurodevelopmental Disorders
Brief Title: Dialogical Family Guidance PostDoc Study
Acronym: DFG II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Diana Cavonius-Rintahaka, PhD, Tampere University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HUS/7626/2023
Record Dates: First submitted 2024-03-07; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Family Dynamics; Family Relations; Family Support
Keywords: neurodevelopmental disorders; family health; family functionality; family support
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Families attending the study Group I: receives Dialogical Family Guidance intervention and they fill questionnaires before and after the intervention.
  Group II: Families do not receive Dialogical Family Guidance (but belong to the same focus group)
Who Masked: Participant, Care Provider
Masking Description: Families include both parents and children. Parents fill the questionnaires, but all family members attend on the meetings during the intervention (six meetings).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): These families receive Dialogical family guidance, including six meetings (during 3 months) within the intervention manual proceedings. Parents fill the questionnaires before and after the intervention.
  Interventions: Behavioral: Dialogical Family Guidance (DFG)
- comparative group (No Intervention): These families (parents in the family) give responses how they manage in ordinary life with their child with neurodevelopmental disorders.
  These families do not receive the intervention.

INTERVENTIONS:
Behavioral: Dialogical Family Guidance (DFG) — DFG is family intervention including six meetings with family members. The individual needs and questions of each family are discussed and issues parents bring up are seemed as important.
  Arms: Intervention group

SUMMARY:
This new family intervention, called Dialogical Family Guidance (DFG) is developed to target family needs especially in families with a child with neurodevelopmental disorders. PhD study showed, that this intervention is functioning with this target group. Participants (families) experienced that they got information, guidance to ordinary life and that the DFG-therapists were listening to them and above all, helping with individual problems and questions. DFG include six meetings and professionals need to attend on a 3-day long education before using this intervention.

DETAILED DESCRIPTION:
Previous studies have highlighted the need for families with a child with neurodevelopmental disorders, to get guidance to daily life, information and also professionals who allow parents to share their own experiences, feelings and questions. Dialogical Family Guidance is developed to offer target families (participants) the help mentioned above. This study is a postdoctoral study to achieve more knowledge and understanding about DFG intervention. This Postdoctoral study is focusing on DFG effectivity offered to families with young children (5-7years). Researchers also want to receive information about DFG effectivity between different units inside and outside the university hospital. Comparation between different units using DFG is one goal with this postdoc study. These results may give researchers deeper understanding when deciding where (university hospital och basic level units) and for whom (childrens age?) DFG intervention is giving the most optimal help.

ELIGIBILITY:
Inclusion Criteria:

* Families with a child with clinical diagnosis within neurodevelopmental ambrella (ADHD, Tourette, Autism disorder, OCD...).
* the child must be between 4-13 years.

Exclusion Criteria:

* Families who do not understand finnish language (because they can not fill the questionnaires and professionals offering DFG are all finnish speaking). At least one parent needs to talk finnish.
* Families who are not motivated to receive DFG.
* Families who do not have a child with neurodevelopmental disorders.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
FAFHES | 0 months and 3 months
  FAFHES (Family Function, Health, and Social Support-questionnaire). The name of the questionnaire explains the content of this questionnaire that includes three sections: family functionality (19 items), family health (23 items), family support provided by professionals (21 items). Likert scale is used with ranging from 1-6 (1= disagree totally......6=I agree totally).

SECONDARY OUTCOMES:
DFG-questionnaire | 3 months
  This questionnaire has been developed for DFG intervention including questions about the intervention sessions and themes. Items are included: e.g. questions about the amount and time consumed on DFG, content as a whole, practical advances, did your family get help, would you recommend this to other families. Likert scale from 1-5 is used. Two open ended questions in the end of the questionnaire is included.
SDQ-p questionnaire (Strengths and difficulties regarding the child) | 0 months and 3 months
  Measures changes in child's behavior. Includes 25 items with 3 point likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Cavonius-Rintahaka, PhD, Principal Investigator — Tampere University, Finland
Locations (1):
- Helsinki university hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
No information is shared regarding the families attending the study. Analyzed study results are shared by using results from scientific study protocols published in academic and international publications.